CLINICAL TRIAL: NCT00256984
Title: A Multi-center Study to Assess the Outcomes of Stapled Trans-Anal Rectal Resection (STARR) in the Treatment of Obstructed Defecation Syndrome (ODS)
Brief Title: Study of Stapled Transanal Rectal Resection (STARR) Surgery in Refractory Constipation Associated With Obstructive Defecation Syndrome (ODS)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ethicon Endo-Surgery (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CI-05-0004
Record Dates: First submitted 2005-11-18; First posted 2005-11-22 (Estimated); Results first posted 2011-04-07 (Estimated); Last update posted 2018-07-16 (Actual); Status verified 2017-10

CONDITIONS: Obstructive Defecation Syndrome; Chronic Constipation; Rectocele; Intussusception
Keywords: Obstructive Defecation Syndrome; Colorectal Surgery; Defecography; Constipation; Rectocele; Intussusception; Quality of Life
MeSH Terms: conditions — Rectocele; Intussusception; Constipation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Stapled Transanal Resection (STARR) with Transtar (PROXIMATE®) 33 mm Circular Stapler

SUMMARY:
The primary purpose of this study is to determine how effective and how durable STARR (stapled transanal rectal resection) surgery is in relieving symptoms of intractable constipation associated with obstructive defecation syndrome (ODS).

DETAILED DESCRIPTION:
Rectocele and rectal intussusception are frequent findings in women but are often asymptomatic apart from anatomical defects, which can be seen on vaginal examination. They can be associated, however, with refractory constipation that may be best described by the terms "Outlet Obstruction" or "Obstructive Defecation Syndrome (ODS)". ODS is characterized by a symptom complex, including the feeling of incomplete evacuation associated with the need to strain excessively and for external assistance (digital, mechanical or positional maneuvers, enemas or suppositories) to aid defecation. Abdominal or rectal pain is also a common complaint. Obstetric trauma is also recognized as a contributing factor. However, none of these symptoms/factors can be singled out to be pathognomonic for this problem. ODS has a prevalence of approximately 12% in the general population.

For individuals with ODS and related intussusception/rectocele, a variety of surgical techniques including abdominal, vaginal, transanal and perineal approaches have been devised. The impact of clinical studies to evaluate these techniques has been limited by variability of results and lack of comparators. Recently, a new surgical approach was developed by an Italian surgeon, A. Longo, and has been evaluated in several European centers. These early studies and observations indicate that this new procedure may in fact provide significantly better symptom resolution in ODS patients than other available treatments, and warrants further study. The procedure is referred to as "Stapled Transanal Rectal Resection (STARR)" and this study will assess its effectiveness in a United States population.

ELIGIBILITY:
Inclusion Criteria:

* Able to comprehend, understand, and speak the English language
* Able to comprehend, follow, and sign an informed consent document (ICD)
* Able to tolerate general or spinal anesthetic
* Often experience excessive straining, sense of incomplete evacuation, and/or prolonged time for complete evacuation when attempting a bowel movement
* Have experienced ODS symptoms for at least 12 months prior to enrollment
* Have a minimum ODS score of 10
* Have rectocele and/or rectal intussusception confirmed by defecography
* Screened for colorectal neoplasia within 7 years of the screening visit (e.g., colonoscopy or barium enema)
* Have an American Society of Anesthesiologists (ASA) score of no more than 3
* Willing to comply with evaluation and management schedule through 5-year follow-up

Exclusion Criteria:

* Fecal incontinence to solid stool
* Full-thickness prolapse
* Perineal infection
* Recto-vaginal fistula
* Enterocele (at rest)
* Any complex pelvic floor prolapse requiring a combined surgical approach
* Prior sigmoid or anterior resection or prior rectal anastomosis
* Presence of foreign material adjacent to the rectum (e.g., vaginal mesh)
* Grade IV hemorrhoids
* Pregnancy
* Chronic narcotic use
* Evidence of colorectal neoplasia, carcinoma, or inflammatory bowel disease
* Physical or psychological condition which would impair study participation
* Unable or unwilling to attend follow-up visits and examinations
* Surgical procedure required concurrently with STARR
* Prior pelvic radiotherapy
* Failure to identify any anatomical or physiological abnormality in the evaluation
* Significant rectal fibrosis
* Anal stenosis precluding insertion of the stapling device
* Participation in any other investigational device or drug study 30 days prior to enrollment
* Presence or history of hepatitis B, hepatitis C, and/or HIV positive test

Ages: 21 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2005-10-01 (Actual); Primary Completion 2008-03-01 (Actual); Study Completion 2008-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robin F Scamuffa, MS, Study Director — Ethicon Endo-Surgery; William Bernie, MD, Study Director — Ethicon Endo-Surgery; Anthony J Senagore, MD, Principal Investigator — Medical University of Ohio; Anders F Mellgren, MD, PhD, Principal Investigator — University of Minnesota
Locations (7):
- United States (7):
  - Colon and Rectal Clinic of Orlando, Orlando, Florida
  - Lahey Clinic, Burlington, Massachusetts
  - Colon & Rectal Surgery Associates Ltd., Minneapolis, Minnesota
  - University Hospitals of Cleveland, Cleveland, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Medical University of Ohio, Department of Surgery, Toledo, Ohio
  - Portland Medical Center, Portland, Oregon

REFERENCES:
- [Background] Shorvon PJ, McHugh S, Diamant NE, Somers S, Stevenson GW. Defecography in normal volunteers: results and implications. Gut. 1989 Dec;30(12):1737-49. doi: 10.1136/gut.30.12.1737. PMID 2612988
- [Background] Kenton K, Shott S, Brubaker L. The anatomic and functional variability of rectoceles in women. Int Urogynecol J Pelvic Floor Dysfunct. 1999;10(2):96-9. doi: 10.1007/pl00004019. PMID 10384970
- [Background] Talley NJ, Weaver AL, Zinsmeister AR, Melton LJ 3rd. Functional constipation and outlet delay: a population-based study. Gastroenterology. 1993 Sep;105(3):781-90. doi: 10.1016/0016-5085(93)90896-k. PMID 8359649
- [Background] Siproudhis L, Dautreme S, Ropert A, Briand H, Renet C, Beusnel C, Juguet F, Rabot AF, Bretagne JF, Gosselin M. Anismus and biofeedback: who benefits? Eur J Gastroenterol Hepatol. 1995 Jun;7(6):547-52. PMID 7552638
- [Background] van Dam JH, Hop WC, Schouten WR. Analysis of patients with poor outcome of rectocele repair. Dis Colon Rectum. 2000 Nov;43(11):1556-60. doi: 10.1007/BF02236738. PMID 11089592
- [Background] Fleshman JW, Fry RD, Kodner IJ. The surgical management of constipation. Baillieres Clin Gastroenterol. 1992 Mar;6(1):145-62. doi: 10.1016/0950-3528(92)90024-9. PMID 1586766
- [Background] Altomare DF, Rinaldi M, Veglia A, Petrolino M, De Fazio M, Sallustio P. Combined perineal and endorectal repair of rectocele by circular stapler: a novel surgical technique. Dis Colon Rectum. 2002 Nov;45(11):1549-52. doi: 10.1007/s10350-004-6465-9. PMID 12432306
- [Background] Dodi G, Pietroletti R, Milito G, Binda G, Pescatori M. Bleeding, incontinence, pain and constipation after STARR transanal double stapling rectotomy for obstructed defecation. Tech Coloproctol. 2003 Oct;7(3):148-53. doi: 10.1007/s10151-003-0026-4. PMID 14628157
- [Background] Boccasanta P, Venturi M, Stuto A, Bottini C, Caviglia A, Carriero A, Mascagni D, Mauri R, Sofo L, Landolfi V. Stapled transanal rectal resection for outlet obstruction: a prospective, multicenter trial. Dis Colon Rectum. 2004 Aug;47(8):1285-96; discussion 1296-7. doi: 10.1007/s10350-004-0582-3. PMID 15484341
- [Background] Boccasanta P, Venturi M, Salamina G, Cesana BM, Bernasconi F, Roviaro G. New trends in the surgical treatment of outlet obstruction: clinical and functional results of two novel transanal stapled techniques from a randomised controlled trial. Int J Colorectal Dis. 2004 Jul;19(4):359-69. doi: 10.1007/s00384-003-0572-2. Epub 2004 Mar 13. PMID 15024596
- [Background] Pescatori M, Dodi G, Salafia C, Zbar AP. Rectovaginal fistula after double-stapled transanal rectotomy (STARR) for obstructed defaecation. Int J Colorectal Dis. 2005 Jan;20(1):83-5. doi: 10.1007/s00384-004-0658-5. Epub 2004 Sep 2. No abstract available. PMID 15349740
- [Background] Grassi R, Romano S, Micera O, Fioroni C, Boller B. Radiographic findings of post-operative double stapled trans anal rectal resection (STARR) in patient with obstructed defecation syndrome (ODS). Eur J Radiol. 2005 Mar;53(3):410-6. doi: 10.1016/j.ejrad.2004.12.012. PMID 15741014
- [Background] Mongardini M, Custureri F, Schillaci F, Cola A, Maturo A, Fanello G, Corelli S, Pappalardo G. [Prevention of post-operative pain and haemorrhage in PPH (Procedure for Prolapse and Hemorrhoids) and STARR (Stapled Trans-Anal Rectal Resection). Preliminary results in 261 cases]. G Chir. 2005 Apr;26(4):157-61. Italian. PMID 16035252
- [Background] Binda GA, Pescatori M, Romano G. The dark side of double-stapled transanal rectal resection. Dis Colon Rectum. 2005 Sep;48(9):1830-1; author reply 1831-2. doi: 10.1007/s10350-005-0103-z. No abstract available. PMID 15991070
- [Background] Jayne DG, Finan PJ. Stapled transanal rectal resection for obstructed defaecation and evidence-based practice. Br J Surg. 2005 Jul;92(7):793-4. doi: 10.1002/bjs.5092. No abstract available. PMID 15962257
- [Background] Talley NJ, Phillips SF, Wiltgen CM, Zinsmeister AR, Melton LJ 3rd. Assessment of functional gastrointestinal disease: the bowel disease questionnaire. Mayo Clin Proc. 1990 Nov;65(11):1456-79. doi: 10.1016/s0025-6196(12)62169-7. PMID 2232900

RESULTS

PARTICIPANT FLOW:
Groups:
- Stapled Trans-Anal Rectal Resection (STARR): STARR procedure (an anterior and posterior, full-thickness stapling and resection of the rectal wall) to correct Obstructive Defecation Syndrome symptoms utilizing the TransStar Circular Stapler
Period: Overall Study
Arm/Group | Stapled Trans-Anal Rectal Resection (STARR)
Started | 75
Completed | 59
Not Completed | 16

BASELINE CHARACTERISTICS:
Arm/Group | Stapled Trans-Anal Rectal Resection (STARR)
Number analyzed (Participants) | 75
Age, Continuous [Median (Full Range); unit: years] — Median age at consent
  years | 48 [23 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75
  Male | 0
ODS composite score [Mean (Standard Deviation); unit: units on a scale] — Based upon Obstructed Defecation Syndrome (ODS) questionnaire. This questionnaire has eight questions, each dealing with frequency of a particular attribute associated with ODS (mechanical, difficulties to evacuate, digitation to evacuate, return to toilet to evacuate, feeling of incomplete evacuation, straining to evacuate, time needed to evacuate, and lifestyle alterations). Each is scored 0-3 (low to high on scale, no units. "0" is the lowest frequency of occurrence, "3" is the highest frequency of occurrence; the total of all attributes (0-24) is the final score.
  units on a scale | 6.19 (3.13)
number of subjects in each age range having STARR procedure [Number; unit: participants]
  <=29 years | 4
  Between 30 and 39 years | 9
  Between 40 and 49 years | 26
  Between 50 and 59 years | 18
  Between 60 and 69 years | 11
  >=70 years | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Change (Reduction) in Total ODS Symptom Composite Score From Baseline to One Year Post Procedure
Description: The primary endpoint used to assess effectiveness of STARR for treatment of ODS was the percentage of change in total ODS symptom composite score (0=worst, 24=best) 1 year after completion of the procedure.
Time Frame: one year from Baseline
Population: Per protocol
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Stapled Trans-Anal Rectal Resection (STARR)
Number analyzed (Participants) | 59
percentage of change | 60.8 (35.46)

2. Secondary Outcome: Percentage of Change in ODS Symptom Composite Score From Baseline at 1 Month Post Procedure
Description: Percentage of change in Obstructive Defecation Syndrome (ODS) symptom composite score from baseline at 1 month post procedure. This score is based on a series of questions designed to understand the extent ODS effects an individual's daily lifestyle (0 is worst score, 24 is best score). Sizing consistent with primary outcome; analysis was per-protocol.
Time Frame: Baseline, 1 month post procedure
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Stapled Trans-Anal Rectal Resection (STARR)
Number analyzed (Participants) | 59
percentage of change | -50.7 (34.4)

3. Secondary Outcome: Maximum Change in Subject-reported Assessment of Symptom Severity and Frequency (PAC SYM).
Description: Assessed as patient-reported assessment of symptom severity and frequency (PAC-SYM)associated with constipation. Patient response options are absent, mild, moderate, severe, and very severe.12 questions relate to severity, 8 questions relate to frequency of symptoms. The lower the score, the less severe the symptoms. Sizing consistent with primary outcome; analysis was per-protocol.
Time Frame: Baseline, 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stapled Trans-Anal Rectal Resection (STARR)
Number analyzed (Participants) | 59
units on a scale | 1.43 (0.72)

4. Secondary Outcome: Percentage of Change in ODS Symptom Composite Score From Baseline at 6 Months (0 is Worst Score, 24 is Best Score)
Description: as for outcome 1
Time Frame: Baseline, 6 months post procedure
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Stapled Trans-Anal Rectal Resection (STARR)
Number analyzed (Participants) | 59
percentage of change | -57.0 (34.4)

5. Secondary Outcome: PAC QOL Patient Assessment of Constipation (Overall)
Description: PAC-QOL is Patient Assessment of Constipation, Quality of Life. The instrument consists of 28 questions on a 0-4 scale. A lower score indicates better quality of life. The score is a number without units.Change from baseline in patient assessment of constipation in quality of life as measured by the PAC QOL instrument score. The questions are designed to measure the impact constipation has had on daily life during the week prior to the subject visit. Sizing was consistent with the primary outcome; analysis was per-protocol
Time Frame: Baseline, 12 months
Population: Sizing consistent with primary outcome; analysis was Intent-to-Treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stapled Trans-Anal Rectal Resection (STARR)
Number analyzed (Participants) | 59
units on a scale | 0.95 (0.996)

6. Secondary Outcome: SF-12 QOL Change From Baseline (Physical Component)at 12 Months
Description: The SF-12 is a validated 12 question quality-of-life questionnaire. The SF-12 extracts 12 items from the SF-36 questionnaire in two six-item subscales, PCS (physical functioning) and MCS (emotional functioning). The SF-12 scores can range from 10 (maximum impairment) to 70 (no impairment). For this study, the endpoint is the percentage of change from baseline over 12 months post procedure.
Time Frame: Baseline, 12 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stapled Trans-Anal Rectal Resection (STARR)
Number analyzed (Participants) | 59
units on a scale | 6.32 (9.106)

7. Secondary Outcome: SF-12 QOL Change (Mental Component) at 12 Months From Baseline
Description: SF 12 change from baseline, mental component. The SF-12 is a validated 12 question quality-of-life questionnaire. The SF-12 extracts 12 items from the SF-36 questionnaire in two six-item subscales, PCS (physical functioning) and MCS (emotional functioning). The SF-36 scores range from 0 (maximum impairment) to 100 (no impairment), the SF-12 scores range from 10 (maximum impairment) to 70 (no impairment). For this study, the endpoint is the percentage of change from baseline over 12 months post procedure.
Time Frame: Baseline, 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stapled Trans-Anal Rectal Resection (STARR)
Number analyzed (Participants) | 59
units on a scale | 4.83 (11.67)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Stapled Trans-Anal Rectal Resection (STARR)
Serious Adverse Events (participants affected / at risk) | 14/75
Other Adverse Events (participants affected / at risk) | 33/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stapled Trans-Anal Rectal Resection (STARR) (N=75)
Blood count abnormal (Investigations) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colostomy (Surgical and medical procedures) | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1
Gastroenteritis (Infections and infestations) | 1
Gastrointestinal injury (Injury, poisoning and procedural complications) | 1
Haematoma infection (Infections and infestations) | 1
Intestinal hypomotility (Gastrointestinal disorders) | 1
Postprocedural haemorrhage (Injury, poisoning and procedural complications) | 2
Rectal haemorrhage (Gastrointestinal disorders) | 1
Rectal perforation (Gastrointestinal disorders) | 1
Suture related complication (Injury, poisoning and procedural complications) | 1
Umbilical hernia (Gastrointestinal disorders) | 1
Urinary retention (Renal and urinary disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stapled Trans-Anal Rectal Resection (STARR) (N=75)
Dizziness (Nervous system disorders) | 6
Insomnia (Psychiatric disorders) | 7
Pruritus (Skin and subcutaneous tissue disorders) | 6
urinary retention (Renal and urinary disorders) | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less